CLINICAL TRIAL: NCT02936687
Title: Mechanisms of Cerebrovascular Control: Acute Insulin Surges Lead to Brain Hypoperfusion in Human Metabolic Syndrome
Brief Title: Mechanisms of Cerebrovascular Control
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: American Heart Association (Other); American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-0197; A176000 (Other: UW Madison); EDUC\KINESIOLOGY\KINESIO (Other: UW Madison); 1-16-ICTS-099 (Other Grant/Funding Number: American Diabetes Association); 15POST23100020 (Other Grant/Funding Number: American Heart Association); Protocol Version 9/3/2020 (Other: UW Madison)
Record Dates: First submitted 2016-09-28; First posted 2016-10-18 (Estimated); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Metabolic Syndrome X
Keywords: blood flow; magnetic resonance imaging; insulin; vasodilation
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Aneurysm | interventions — omega-N-Methylarginine; ambrisentan; Sodium Chloride; Vascular Access Devices; Glucose Tolerance Test; Lactose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Metabolic Syndrome NOS Inhibition (Experimental): Will occur over two separate study visits after screening. Eligible subjects with MetSyn will undergo NOS Inhibition during one visit and placebo infusion in the other visit. Subjects will also undergo 3 Tesla MRI scanning and an intravenous catheter, and will complete an Oral Glucose Tolerance Test during the study visits. More details under Study Description.
  Interventions: Drug: NOS Inhibition; Drug: NOS Inhibition Placebo; Device: 3 Tesla MRI; Device: Intravenous Catheter; Other: Oral Glucose Tolerance Test
- Metabolic Syndrome ET-1 Inhibition (Experimental): Will occur over two separate study visits after screening. Eligible male subjects with MetSyn will complete an oral ET-1 Inhibition during one visit and an oral placebo in the other visit. Subjects will also undergo 3 Tesla MRI scanning and an intravenous catheter, and will complete an Oral Glucose Tolerance Test during the study visits. More details under Study Description.
  Interventions: Drug: ET-1 Inhibition; Device: 3 Tesla MRI; Device: Intravenous Catheter; Other: Oral Glucose Tolerance Test; Drug: ET-1 Inhibition Placebo
- Control NOS Inhibition (Experimental): Will occur over two separate study visits after screening. Eligible control subjects will undergo NOS Inhibition during one visit and placebo infusion in the other visit. Subjects will also undergo 3 Tesla MRI scanning and an intravenous catheter, and will complete an Oral Glucose Tolerance Test during the study visits. More details under Study Description.
  Interventions: Drug: NOS Inhibition; Drug: NOS Inhibition Placebo; Device: 3 Tesla MRI; Device: Intravenous Catheter; Other: Oral Glucose Tolerance Test
- Control ET-1 Inhibition (Experimental): Will occur over two separate study visits after screening. Eligible male control subjects will complete an oral ET-1 Inhibition during one visit and an oral placebo in the other visit. Subjects will also undergo 3 Tesla MRI scanning and an intravenous catheter, and will complete an Oral Glucose Tolerance Test during the study visits. More details under Study Description.
  Interventions: Drug: ET-1 Inhibition; Device: 3 Tesla MRI; Device: Intravenous Catheter; Other: Oral Glucose Tolerance Test; Drug: ET-1 Inhibition Placebo

INTERVENTIONS:
Drug: NOS Inhibition — NOS inhibition: L - NMMA is a potent non-selective NOS inhibitor used to study vascular physiology. L-NMMA will be infused at 3 mg/kg body weight/hr bolus (over 10min ) followed by a maintenance infusion of 1 mg/kg/hr for the duration of the experiment. Systemic delivery of L - NMMA has been shown to elevate blood pressure ~8-15 mmHg that is within the range observed during exercise.
  Other Names: L-NMMA
  Arms: Control NOS Inhibition; Metabolic Syndrome NOS Inhibition
Drug: ET-1 Inhibition — ET-1 inhibition: Ambrisentan is an antagonist of the ETA receptor. Subjects will receive 10 mg of Ambrisentan in a pill form 90-150 minutes prior to the OGTT. This class of drugs have been used to research ET-1 signaling in diabetes, obesity, and hypertension. ETA receptors are the most likely to mediate excessive constriction in MetSyn patients. Ambrisentan will be taken orally. Systemic delivery of endothelin antagonist have been shown at chronic dosing to decrease systolic blood pressure 4.5±10 mmHg and diastolic 3 ± 7.5 mmHg in hypertensives, and not alter mean arterial pressure in obesity.
  Other Names: Ambrisentan
  Arms: Control ET-1 Inhibition; Metabolic Syndrome ET-1 Inhibition
Drug: NOS Inhibition Placebo — Saline will be infused at the same rate and quantity as the corresponding drug visit.
  Other Names: Saline
  Arms: Control NOS Inhibition; Metabolic Syndrome NOS Inhibition
Device: 3 Tesla MRI — A 3 Tesla MRI will be used to quantify cerebral blood flow and capture cerebral vessel structure at designated time points throughout the study visits (at baseline and during treatment conditions).
  Other Names: MRI
Device: Intravenous Catheter — A blood sampling IV catheter will be used to draw up to 15 mL blood samples at specific time points throughout each study visit to measure concentrations of glucose and insulin as well as for markers of inflammation and oxidative stress.
  Other Names: Cath
Other: Oral Glucose Tolerance Test — The subject will drink distilled deionized water (300ml) containing 75 grams glucose within 5 minutes.
  Other Names: OGTT
Drug: ET-1 Inhibition Placebo — Placebo pill similar in size and shape to Ambrisentan will be used as placebo control.
  Other Names: Lactose Capsules
  Arms: Control ET-1 Inhibition; Metabolic Syndrome ET-1 Inhibition

SUMMARY:
The objective of this study is to identify insulin-specific cerebral blood flow (CBF) control mechanisms, and establish cerebrovascular responsive baseline in younger (18-45 yrs) metabolic syndrome adults (MetSyn) who are at substantial risk of stroke and other types of cardiovascular mortality even if they never develop diabetes. The central hypothesis is that vasodilator actions of insulin are impaired in MetSyn due to loss of dilator and gain of constrictor signals. This study will focus on 2 mechanisms that likely limit CBF in MetSyn: 1) Disruption of nitric oxide (NO) vasodilation, and 2) Exaggerated endothelin (ET-1) constriction. Three specific aims will be addressed: Aim 1: To test the hypothesis that physiologic surges of insulin acutely increase CBF in young adults, but adults with MetSyn exhibit paradoxical insulin-mediated vasoconstriction. Aim 2: To test the hypotheses that key mechanisms responsible for poor CBF in MetSyn are shifts in NO and ET-1 signaling. Specifically, in healthy controls, NO mediates robust dilation, with little to no ET-1 constriction. In contrast, adults with MetSyn exhibit uncoupled NO synthase (NOS) and exaggerated ET-1 constriction. Aim 3: To test the hypothesis that insulin regulation of CBF is regionally distinct (e.g. Middle Cerebral Artery (MCA) reactive than Anterior Cerebral Artery (ACA) or basilar), and the negative effects of insulin resistance (IR) are similarly regionally specific.

DETAILED DESCRIPTION:
Introduction It is widely accepted that insulin resistance in MetSyn increases the risk of cerebrovascular disease (CVD) and stroke. Additionally, MetSyn is associated with cognitive impairments and increased risk of neurodegenerative diseases. Despite strong association of poor cerebrovascular health in MetSyn, the cerebral blood flow (CBF) response to acute insulin surges in humans remains largely unexplored. Cerebrovascular dysfunction in response to insulin and potential mechanism(s) that attenuate CBF may not only highlight the central underpinnings of the pathophysiology of stroke and CVD, it may provide key insights to understanding cognitive decline strongly linked to older individuals with MetSyn. Therefore, establishing the mechanisms of insulin-mediated cerebrovascular control are not only important for decreasing mortality in MetSyn, it may be profoundly important to maintaining brain health. Insulin-meditated vasodilation is largely a vascular endothelium-dependent process. Elegant experiments using animal models suggests insulin resistance disrupts six endothelial signaling pathways, with the strongest evidence implicating a loss of nitric oxide (NO) vasodilation, and exaggerated endothelin (ET-1) constriction. The literature indicates that in MetSyn, a spike in insulin leads to vasoconstriction and cerebral hypoperfusion. These findings are directionally opposite from no change or insulin-mediated vasodilation and increase in CBF reported in the literature. Evidence suggests that uncoupled function of nitric oxide synthase (NOS) leads to unfavorable balance between NO, reactive oxygen species, and ET-1. Normally, stimulation of insulin receptor on the vascular endothelium should provide an environment in which NOS manufactures NO leading to vasodilation and inhibition of ET-1. Instead, in MetSyn insulin stimulates the vasoconstrictor ET-1 to a greater extent while, NOS is uncoupled generating more reactive oxygen species that scavenges the NO that is generated leading to a greater vasoconstrictor signal rather than vasodilation.

Specific Aims/Study Objectives

Specific Aims:

The central hypothesis is that vasodilator actions of insulin are already impaired in metabolic syndrome due to loss of dilator and gain of constrictor signals. Cerebral vasodilation to insulin is largely endothelium-dependent. Emerging evidence in animal models suggests insulin resistance disrupts at least six endothelial signaling pathways that could be potential targets, and this proposal focuses on two that most likely reduce CBF in MetSyn: 1) Loss of nitric oxide (NO) vasodilation, and 2) Exaggerated endothelin (ET-1) constriction. These experiments will address three specific aims:

Aim 1: To test the hypothesis that physiologic surges of insulin acutely increase CBF in young adults, but adults with MetSyn exhibit paradoxical insulin-mediated vasoconstriction.

Aim 2: To test the hypotheses that key mechanisms responsible for poor CBF in MetSyn are shifts in NO and ET-1 signaling. Specifically, in healthy controls, NO mediates robust dilation, with little to no ET-1 constriction. In contrast, adults with MetSyn exhibit uncoupled NO synthase (NOS) and exaggerated ET-1 constriction.

Aim 3: To test the hypothesis that insulin regulation of CBF is regionally distinct (e.g. MCA reactive than ACA or basilar), and the negative effects of IR are similarly regionally specific.

Hypotheses:

* Adults with metabolic syndrome will exhibit reduced cerebral vasodilation in response to an OGTT
* NOS inhibition will reduce the CBF responses (Δ CVC/Δ insulin) in lean controls to levels of Metabolic syndrome whereas it will increase CBF responses in Metabolic syndrome, suggesting that Metabolic syndrome have uncoupled NOS function
* ET-1 inhibition will increase CBF responses (Δ Cerebral Vascular Conductance Index (CVCi)/Δ insulin) in lean controls and metabolic syndrome. However, it will increase significantly more in in metabolic syndrome.
* The MCA will be more reactive to insulin surges than other cerebral arteries

Study Endpoints: Change in Cerebral vascular conductance (CVC, ml/min/100mmHg) relative to the change in concentration of insulin in blood after consumption of glucose.

Subjects Sixty participants (30 per group) will be recruited. Determination of eligibility will be a two-step process. The first step is all participants will complete an initial screen to determine if they qualify for the screening visit. Preliminary eligible subjects will be invited to the research lab for informed consent and formal screening.

During the screening visit at the research laboratory, subjects will complete informed consent, a health history questionnaire, an MRI Safety screening form, and a physical activity questionnaire. Height, weight, blood pressure, and waist and hip circumference will also be taken. Additionally, a venous blood sample will be drawn for glucose and lipid testing to determine eligibility. If the screening visit reveals that there is an abnormality or contraindication to participation, which is covered or not covered in the summarized exclusion criteria, the potential subject will not be allowed to participate. As a summary, subjects will experience the following activities during the in-lab screening visit:

Methods Following initial screening and a screening visit, participation in this study will involve two separate MRI study visits (Saline infusion as placebo, versus L-NMMA infusion to inhibit NOS OR Ambrisentan orally (male participants only), versus Lactose placebo orally to inhibit ET-1). Subjects will be directed into an experimental condition (placebo/L-NMMA or placebo/Ambrisentan) based on number of subjects need to maintain statistical power. For the Ambrisentan trial, subjects must be male, due to potential harmful effects of drug on fetus. Once assigned an experimental condition group, the drug order (placebo/drug) will be performed in a randomly assigned, counter-balanced single blind fashion. The experimental procedures will be identical on all testing days with the exception of which drug will be infused. Throughout each visit, subjects will be monitored for heart rate, blood pressure, end-tidal carbon dioxide, and verbal communication of adverse symptoms (how is the subject feeling) while in the MRI scanner.

Pregnancy Test: All female subjects must have a negative urine pregnancy test prior to either study visits (placebo or drug) to ensure they are not pregnant at the time of each study visit. Females will not be assigned to the Ambrisentan trial, even if their pregnancy test is negative.

Venipuncture Blood Sample: During the screening visit, blood (up to 20 ml) will be drawn using venipuncture to be analyzed for fasting glucose, serum lipids.

Subjects will abstain from exercise, caffeine, and NSAIDS, as well as fast for ≥ 10 hours prior to all experimental trials.

Intravenous Catheter: Trained staff will place two intravenous catheters. Placement of the catheters will be in any arm veins deemed most suitable for ease of access. However, one will be placed in the antecubital fossa (infusion), and one in the antecubital, hand, or wrist vein (blood sample) of the opposite arm for each of the two study visits. The blood sampling IV catheter will be used to draw up to 15 mL blood samples at specific time points throughout each study visit to measure concentrations of glucose and insulin as well as for markers of inflammation and oxidative stress. All procedures are identical during each trial (placebo/L-NMMA/BQ123). The specific time points, which are approximate due to small variations in MRI scan times, are as follows:

* Baseline, prior to baseline PC VIPR scan
* Before PC VIPR scan 1 after OGTT
* Before PC VIPR scan 2 after OGTT
* Before PC VIPR scan 3 after OGTT
* Before PC VIPR scan 4 after OGTT
* Before PC VIPR scan 5 after OGTT
* Before PC VIPR scan 6 after OGTT
* Before PC VIPR scan 7 after OGTT
* Before PC VIPR scan 8 after OGTT
* Before PC VIPR scan 9 after OGTT

Intra-venous infusion:

I. NOS inhibition: L - NMMA is a potent non-selective NOS inhibitor used to study vascular physiology. L-NMMA will be infused at 3 mg/kg body weight/hr bolus (over 10min ) followed by a maintenance infusion of 1 mg/kg/hr for the duration of the experiment. Systemic delivery of L - NMMA has been shown to elevate blood pressure ~8-15 mmHg that is within the range observed during exercise.

II. Placebo: Placebo infusion rates will be determined using the same formulas for L-NMMA infusion, using the subject's most recent screening weight. Ideally, saline will be infused at the same rate and quantity as the corresponding drug visit. Subject's that are rescreened and have a weight change, however, may have a saline infusion rate that differs slightly from the L-NMMA infusion rate.

A small discrepancy in saline and drug infusion rate is insignificant from a scientific perspective as there is already variability in the amount of saline that the subject receives since it is used to flush the IV (1-5 mL) with every blood draw (up to 10 blood draws).

ET-1 - Inhibition studies (15 control, 15 MetSyn) (Ambrisentan Arm):

I. ET-1 inhibition: Ambrisentan is an antagonist of the ETA receptor. Subjects will receive 10 mg of Ambrisentan in a pill form 90-150 minutes prior to the OGTT. This class of drugs have been used to research ET-1 signaling in diabetes, obesity, and hypertension (Bruno, Sudano, Ghiadoni, Masi, & Taddei, 2010; Lteif, Vaishnava, Baron, & Mather, 2007; Mather, Mirzamohammadi, Lteif, Steinberg, & Baron, 2002). ETA receptors are the most likely to mediate excessive constriction in MetSyn patients. Ambrisentan will be taken orally. Systemic delivery of endothelin antagonist have been shown at chronic dosing to decrease systolic blood pressure 4.5±10 mmHg and diastolic 3 ± 7.5 mmHg in hypertensives, and not alter mean arterial pressure in obesity (Bruno et al., 2010; Mather et al., 2010; Spratt et al., 2001).

II. Placebo: Placebo pill similar in size and shape to Ambrisentan will be used as placebo control.

Magnetic Resonance Imaging (MRI): A 3 Tesla MRI will be used to quantify cerebral blood flow and capture cerebral vessel structure at designated time points throughout the study visits (at baseline and during treatment conditions). No contrast agent will be used at any time. The subject will be in the scanner for an initial baseline scan and during the experimental trials. All scanning will be accomplished in the proposed timeline of experimental trials. While in the scanner, subjects will be monitored for heart rate, ECG, end-tidal carbon dioxide (CO2), and blood pressure. The scanner has the capabilities to collect this data, except for end-tidal CO2, which will be collected with a subject monitor. In addition to standard pulse sequences commonly obtained for clinical purposes (localizers, standard MR Angiography for vessel anatomy (without a contrast agent), 2D phase contrast MRI for velocity encoded measurements), a.s.o.; 'basic sequences'), an acquisition scheme developed at the University of Wisconsin-Madison will be used. This scheme, PC VIPR (phase contrast vastly under-sampled isotropic projection reconstruction) is unique in its capability to acquire volumetric data sets with three-directional velocity encoding and high spatial resolution in fairly short scan times. All pulse sequences used in this study are designed to stay within the current guidelines for dB/dt established by the FDA.

Oral Glucose Tolerance Test (OGTT): The subject will drink distilled deionized water (300ml) containing 75 grams glucose within 5 minutes. This is the standard administration of OGTT.

Re-enrollment: Male subjects that fully complete the study will have the choice to re-enroll and complete the wing of the study they did not participate in. Subjects will be re-screened to determine eligibility and will be separated by at least 1 week from completion of the study. Furthermore, they only participate in the L-NMMA or Ambrisentan (which ever they have not completed in the other wing of the study), they will not need to repeat the control/saline visit.

ELIGIBILITY:
* Inclusion Criteria (all):

  * Sedentary (≤ 90 minutes of vigorous physical activity per week)
  * Women must be premenopausal with a regular menstrual cycle
  * For the Ambrisentan trial, participants must be male, due to potential harmful effects of drug on fetus
* Inclusion Criteria (Controls):

  * Participants will be lean (BMI ≥19 - ≤25 kg/m2)
  * Sedentary (≤ 90 minutes of vigorous physical activity per week)
  * Without any cardiovascular co-morbidities
* Inclusion Criteria: (Metabolic Syndrome):

  * Participants must qualify under the National Cholesterol Education Program-Adult Treatment Panel III (NCEP-ATP III) definition of metabolic syndrome as modified by the American Heart Association and International Diabetes Federation. Participants must meet 3 or more of the following 5 criteria:

    * fasting glucose ≥ 100 mg/dL,
    * fasting triglycerides ≥ 150 mg/dL,
    * elevated blood pressure (≥ 130 systolic and/or ≥ 85 diastolic mmHg),
    * waist circumference at the iliac crest > 102 cm (men) or ≥ 88 cm (women).
* Exclusion Criteria:

  * Fasting glucose ≥ 126 mg/dL
  * Having ≥1- ≤ 2 of the above criteria for MetSyn.
  * Personal medical history of coronary artery disease, stroke, heart attack, heart valve disease, congestive heart failure, previous heart surgery, history of lung disease (Note: asthma that is not currently active and being treated is NOT considered an exclusion criteria) or peripheral artery disease, or history of renal/kidney and liver/hepatic disease.
  * Taking metabolic medications (insulin-sensitizing, lipid-lowering medications, etc.) or any medications for cardiovascular-related issues will be excluded.
  * Current use of tobacco (i.e. smoke, smokeless, and vapor). If participant has used tobacco products ≤10 in the last year and ≤1 time in the last month, he or she will still be considered eligible.
  * Females will be excluded if pregnant, lactating, or postmenopausal.
  * Participants having any contraindications of having an MRI (such as claustrophobia, metallic implant, etc.).
  * Participant has an abnormality or contraindication to study participation, which is not covered in the eligibility criteria.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change in cerebrovascular blood flow in response to NOS inhibition. | Through study completion (an average of 2 years)
  A 3 Tesla MRI will be used to quantify cerebral blood flow and capture cerebral vessel structure at designated time points throughout the study visits.
Change in cerebrovascular blood flow in response to ET-1 inhibition. | Through study completion (an average of 2 years)
  A 3 Tesla MRI will be used to quantify cerebral blood flow and capture cerebral vessel structure at designated time points throughout the study visits.

CONTACTS AND LOCATIONS:
Overall Officials: William G. Schrage, Ph.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No